CLINICAL TRIAL: NCT03465280
Title: Airway Intervention Registry (AIR) Extension: Recurrent Respiratory Papillomatosis
Brief Title: Airway Intervention Registry (AIR): Recurrent Respiratory Papillomatosis (RRP)
Acronym: AIR:RRP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 08733
Record Dates: First submitted 2018-02-26; First posted 2018-03-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Respiratory Papillomatosis; Human Papilloma Virus
Keywords: Recurrent respiratory papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Surgical Instruments; Lasers, Gas; potassium titanylphosphate; Lasers; Lasers, Dye; Radiofrequency Ablation; Acyclovir; artemisinin; Bevacizumab; Celecoxib; Cidofovir; Cimetidine; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; indole-3-carbinol; Interferon-alpha; Methotrexate; Tretinoin; Isotretinoin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 53 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Microdebrider — Removal of lesions via microdebrider
Procedure: Cold-steel surgery (forceps) — Removal of lesions via forceps
Procedure: Carbon dioxide laser — Removal of lesions via carbon dioxide laser
Procedure: Potassium titanyl phosphate (KTP) laser — Removal of lesions via KTP laser
Procedure: Pulsed dye laser — Removal of lesions via pulsed dye laser
Procedure: Radiofrequency ablation — Removal of lesions via radiofrequency ablation
Procedure: Monopolar suction diathermy — Removal of lesions via monopolar suction diathermy
Procedure: Plasma coagulation — Removal of lesions via plasma coagulation
Procedure: Other — Removal of lesions via other methods
Other: Adjuvant therapies — All adjuvant therapies
  Other Names: Acyclovir; Artemisinin; Bevacizumab (Avastin); Celecoxib (Celebrex); Cidofovir; Cimetidine; Di-indolmethane (DIM); Gardasil; Indole-3-carbinol (I3C); alpha-Interferon; PEG-Interferon; Methotrexate; Retinoic acid (isotretinoin); Ribavarin; Other

SUMMARY:
Recurrent Respiratory Papillomatosis (RRP) causes wart-like growths in the airway which can make it difficult to breathe, speak and carry out normal everyday activities. It is a rare condition affecting all ages, but is more common and aggressive in children than in adults, affecting 4 in every 100,000 children. There is no known cure for RRP, but symptoms are checked through regular hospital visits, with multiple therapies or procedures under general anaesthetic needed to remove or shrink the growths which can grow back quickly. The problem is that nobody knows which therapies or procedures work best. Aim: To identify which RRP treatments currently used in National Health Service (NHS) hospitals within the United Kingdom (UK) are the most effective and safest in the short- and long-term. It will also identify which patients respond best to specific treatments, and those who are at higher risk of experiencing a complication after treatment.

Method: Collect information from usual patient care and quality of life questionnaire responses in a secure online database. Participation in this study requires patient/parent/guardian consent. This observational study does not require patients to undergo any additional intervention as part of the research.

DETAILED DESCRIPTION:
Primary aim:

The overall goal is to improve the care of patients with Recurrent Respiratory Papillomatosis (RRP) - and the investigators aim to do this by determining the most effective and safe RRP treatments currently being used in patients in National Health Service (NHS) hospitals within the United Kingdom (UK) (information which is currently lacking).

By determining the most effective treatments of RRP, the investigators will be able to increase the time interval between surgical interventions to maintain symptomatic control, reduce overall number of RRP interventions, severity and spread of papillomas in the airway, hospital visits, medications and ultimately improve quality of life in those suffering from RRP. By also capturing peri- and post-procedural details the investigators will be able to determine the relative safety of treatments and identify those which slow the progression of disease.

From the data collected the investigators intend to identify patient subgroups (based on patient characteristics such as age, gender, human papillomavirus (HPV) type, location of papillomas, RRP severity and spread, comorbidities) who respond better to specific treatments, and also identify patient risk factors which contribute to the complication outcomes (such as tracheostomy).

Secondary aims:

* build an evidence base of the different RRP treatments used across the UK which will help to formulate hypotheses for future research in RRP and improve quality of life for RRP patients;
* inform National Institute for Health and Care Excellence (NICE) interventional procedure guidance on radiofrequency cold ablation (IPG434,2012), which is currently under special arrangements due to lack of safety and efficacy evidence;
* identify common symptoms or signs associated with RRP disease profile, to aid future diagnosis of RRP;
* determine the geographical spread of RRP patients across the UK, to inform effective use of future NHS resources and inform the Department of Health strategy in its quadrivalent HPV vaccination programme (protecting against four types of HPV including types 6 and 11 commonly associated with RRP) currently offered to 12-13 year old girls within the NHS childhood vaccination programme;
* inform future development of national clinical guidance on management of RRP to ensure that everyone receives the best care based on best available current knowledge;
* determine impact of COVID on RRP patients including changes to RRP management, RRP symptoms.

Objectives:

The investigators will make use of an existing secure online database platform (the Airway Intervention Registry, AIR - developed and hosted by The Newcastle upon Tyne Hospitals NHS Foundation Trust, NUTH) and its associated infrastructure and develop it to capture additional observational outcomes from standard clinical practice and quality of life questionnaires from RRP patients. All RRP patients (any age) receiving treatment in any UK NHS hospital will be eligible for inclusion. Data collection will be open for 53 months with no minimum follow-up required for patients. Due to its recurrent nature (requiring regular hospital visits to maintain an open airway), following this patient population will allow the investigators to determine both the short- and long-term relative safety and efficacy of RRP treatments used in the UK. Consent will be required (from patients/parent/guardian) before data are entered into the online database.

ELIGIBILITY:
Inclusion Criteria:

* patients of any age (no restrictions) diagnosed with (newly diagnosed or existing) and receiving treatment for respiratory papillomatosis
* informed assent/consent of data participation provided by patient/parent/guardian

Exclusion Criteria:

* patients participating in other studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with respiratory papillomatosis receiving hospital treatment
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Time interval between surgical interventions | Over study duration (53 months)
  Time between surgical interventions to maintain symptomatic control

SECONDARY OUTCOMES:
RRP surgical intervention - nature | Over study duration (53 months)
  Nature of intervention
RRP surgical intervention - timing | Over study duration (53 months)
  Timing of intervention
RRP adjuvant therapy - nature | Over study duration (53 months)
  Nature of intervention
RRP adjuvant therapy - timing | Over study duration (53 months)
  Timing of intervention
Histology results | Over study duration (53 months)
  Including HPV type
Severity of papillomas | Over study duration (53 months)
  Measured via Derkay severity score (higher score corresponding with higher severity; clinical score range 0-11, anatomical score range 0-75, summed total score range 0-86)
Number of hospital visits/attendances | Over study duration (53 months)
  Inpatient, Accident & emergency, Outpatient
Voice assessment (paediatric) | Over study duration (53 months)
  Measured via paediatric voice handicap index (higher score corresponding with higher voice handicap, range 0-99)
Voice assessment (adult) | Over study duration (53 months)
  Measured via voice handicap index (higher score corresponding with higher voice handicap, range 0-120)
Short-term complications | During hospital admission for RRP intervention (length of hospital stay can vary between patients e.g. from 0-100 days)
  Complications arising in-hospital
Post-operative discharge location - planned | During hospital admission for RRP intervention (length of hospital stay can vary between patients e.g. from 0-100 days)
  Planned discharge location (decided pre-operation)
Post-operative discharge location - actual | During hospital admission for RRP intervention (length of hospital stay can vary between patients e.g. from 0-100 days)
  Actual discharge location (occurring post-operation)
Long-term complications | Over study duration (53 months)
  Unexpected hospital, Accident & emergency (A&E), General Practitioner (GP) attendances due to RRP symptoms.
Impact of COVID | From March 2020 onwards (30 months)
  Test results, antibody results, symptoms, changes to management,

CONTACTS AND LOCATIONS:
Overall Officials: Adam Donne, Principal Investigator — Alder Hey Children's NHS Foundation Trust
Locations (48):
- United Kingdom (48):
  - NHS Grampian, Aberdeen
  - Betsi Cadwaladr University Health Board,, Bangor
  - Basildon & Thurrock University Hospitals NHS FT, Basildon
  - Belfast Health and Social Care Trust, Belfast
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospital NHS FT, Blackpool
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Local Health Board, Cardiff
  - North Cumbria Univeristy Hospital NHS Trust, Carlisle
  - Hywel Dda University Health Board, Carmarthen
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh
  - Frimley Health NHS Foundation Trust, Frimley
  - NHS Greater Glasgow & Clyde, Glasgow
  - London North West University Healthcare NHS Trust, Harrow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Great Ormond Street Hospital for Children NHS FT, London
  - Bedfordshire Hospitals NHS Foundation Trust, Luton
  - Manchester University Hospital NHS Foundation Trust, Manchester
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Wirral University Teaching Hospitals NHS Foundation Trust, Metropolitan Borough of Wirral
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Isle of Wight NHS Trust, Newport
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital of Plymouth NHS Trust, Plymouth
  - Swansea Bay University Health Board, Port Talbot
  - East Sussex Healthcare NHS Trust, Saint Leonards-on-Sea
  - Salford Royal NHS Foundation Trust, Salford
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Stockport NHS Foundation Trust, Stockport
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: No
Patients will be informed that all data collected will be used for research purposes, no patient identifiable information will be shared with external parties for commercial purposes, patient identifiable information will only be accessible by clinicians at their treating organisation, pseudonymised data will be accessed by study analysts, and that only anonymised high-level aggregate data will be shared with other centres to update participating centres of study progress and data completeness issues. Patients will also be informed that any external researchers requesting data from the registry will be required to submit a formal application form and evidence of appropriate ethical approvals in place for review by the Steering Group. If approval is given, only anonymised data will be shared for the purposes of external research studies.

REFERENCES:
- [Derived] Donne AJ, Keltie K, Burn J, Belilios E, Powell S, Cognigni P, Nixon IJ, Bateman N, Kubba H, Judd O, Sims A. Current Practice, Safety and Efficacy of Interventions for Recurrent Respiratory Papillomatosis: Evidence From a UK Registry. Clin Otolaryngol. 2025 Mar;50(2):271-279. doi: 10.1111/coa.14245. Epub 2024 Oct 24. PMID 39445512